CLINICAL TRIAL: NCT02767635
Title: Comparison Between Steroid and Two Different Sites of Botulinum Toxin Injection in the Treatment of Lateral Epicondylalgia: A Randomized Double-blind Active Drug-controlled Pilot Study
Brief Title: Comparison Between Steroid and Different Sites of Botulinum Toxin Injection in the Treatment of Lateral Epicondylalgia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Yu-Ching Lin, Visiting Physician, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BR-100-108
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Tennis Elbow
MeSH Terms: conditions — Tennis Elbow | interventions — Botulinum Toxins, Type A; Triamcinolone Acetonide; Steroids

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Botox-Epic group (Experimental): 20 units of Botox injection into lateral epicondyle in Botox-Epic group
  Interventions: Drug: Botox-Epic
- Botox-Tend group (Experimental): 20 units of Botox injected into tender point of muscles in Botox-Tend group
  Interventions: Drug: Botox-Tend
- Steroid group (Active Comparator): 40mg of triamcinolone acetonide but not Botox injected into lateral epicondyle in Steroid group
  Interventions: Drug: triamcinolone acetonide (Steroid)

INTERVENTIONS:
Drug: Botox-Epic — injected 20 units of Botox into lateral epicondyle in Botox-Epic group
  Other Names: onabotulinumtoxinA
  Arms: Botox-Epic group
Drug: Botox-Tend — injected 20 units of Botox into tender point of muscles in Botox-Tend group
  Other Names: onabotulinumtoxinA
  Arms: Botox-Tend group
Drug: triamcinolone acetonide (Steroid) — injected 40mg of triamcinolone acetonide into lateral epicondyle in Steroid group
  Other Names: steroid
  Arms: Steroid group

SUMMARY:
The aim of the study is to compare two different injection sites of low dose botulinum toxin type A with steroid in treating lateral epicondylalgia.

DETAILED DESCRIPTION:
Lateral epicondylalgia or tennis elbow is a common painful elbow disorder with a prevalence of 1% to 3% in the general population and has a higher rate up to 14.5% in strenuous jobs. Botulinum toxin type A injection was an emerging option in treating lateral epicondylalgia. In this study, the patients were randomly assigned into three groups:

1. Botox-Epic group received 20 units of Botox injection into lateral epicondyle;
2. Botox-Tend group had 20 units of Botox injected into tender point of muscles;
3. Steroid group had 40mg of triamcinolone injected into lateral epicondyle.

The aim of this randomized controlled study was to compare the effects of injection with corticosteroid and botulinum toxin type A via two different sites in patients with lateral epicondylalgia.

ELIGIBILITY:
Inclusion Criteria:

* spontaneous local pain over lateral epicondyle of the affected elbow for more than six months and failure to respond to previous physical therapy or oral medications,
* local tenderness around the lateral epicondyle, and
* pain elicited or aggravated by resisted contraction of the wrist or middle finger extensors.

Exclusion Criteria:

* local steroid injection within the past six months,
* coexisting elbow arthritis or arthralgia,
* previous trauma or surgery history over the lateral epicondyle,
* pregnancy or lactation, and
* other systemic, neuromuscular or bleeding disorders that are contraindicated to Botox injection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change of pain assessed on the visual analogue scale | baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks

SECONDARY OUTCOMES:
Change of grip strength by dynamometer | baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks
Change of self-assessment by Patient-Rated Tennis Elbow Evaluation | baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Ching Lin, MD, MSc, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, National Cheng Kung University Hospital, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo YH, Kuan TS, Chen KL, Lien WC, Hsieh PC, Hsieh IC, Chiu SH, Lin YC. Comparison Between Steroid and 2 Different Sites of Botulinum Toxin Injection in the Treatment of Lateral Epicondylalgia: A Randomized, Double-Blind, Active Drug-Controlled Pilot Study. Arch Phys Med Rehabil. 2017 Jan;98(1):36-42. doi: 10.1016/j.apmr.2016.08.475. Epub 2016 Sep 22. PMID 27666156